CLINICAL TRIAL: NCT01202305
Title: The Use of Lymph Node Biopsies to Support HIV Pathogenesis Studies
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-03606
Record Dates: First submitted 2010-09-09; First posted 2010-09-15 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: HIV; HIV persistence; Lymph node fibrosis
MeSH Terms: interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Inguinal LN
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV negative
  Interventions: Procedure: Lymph node biopsy
- HIV positive
  Interventions: Procedure: Lymph node biopsy

INTERVENTIONS:
Procedure: Lymph node biopsy — Inguinal lymph node biopsy

SUMMARY:
HIV medicines have led to dramatic improvements in health. However, there remains a concern for potential drug toxicities, cost of drugs, and need for life-long treatment. In addition, research has found that health is not completely restored in HIV-infected patients, even if they have been taking effective HIV medicines for a long time. This may be due to direct drug-toxicity, continued replication of the virus, and/or inflammation of the body in response to the virus. Therefore, a more complete understanding of how HIV stays in the body is necessary.

Recent research has shown that one of the places that HIV can stay in the body is in lymphatic tissues such as lymph nodes (even in patients who have been taking HIV medicines for a long time). In addition, the amount of damage to the lymphatic tissues can predict how the immune system (CD4+ T cell count) will respond to therapy.

The investigators therefore propose a study in which lymph nodes from the groin area will be removed, with the goals of: 1) seeing how much HIV is in lymph nodes and 2) seeing how much damage has happened to the lymph node architecture.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent
2. No contraindication to surgical procedures
3. Palpable inguinal adenopathy at study entry
4. For HIV seropositive subjects, meeting one of the following criteria: (1) on stable highly active antiretroviral therapy (HAART) with a recent undetectable viral load (< 50 copies/mL) ("HAART suppressed"), (2) antiretroviral untreated with an undetectable viral load (< 50 copies/mL) ("elite" controllers), or (3) antiretroviral untreated with a detectable viral load (> 1000 copies/mL) ("non-controllers")

Exclusion Criteria:

1. Known anemia (HIV+ males Hct<34; females Hct<32) or contraindication to donating blood
2. Blood coagulation disorder (including bleeding tendency or problems in past with blood clots)
3. Platelets < 50,000/mm3
4. PTT > 2x ULN
5. INR > 1.5
6. Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We propose a study in which inguinal lymph node biopsies will be performed on HIV-infected and uninfected subjects, with the goals of: 1) quantifying and characterizing residual virus in lymph nodes and 2) quantifying and comparing lymph node architecture in untreated subjects, HAART-suppressed subjects, elite controllers, and HIV-negative subjects. This research study will permit a lymph node biopsy to be performed and peripheral blood to be obtained from patients with HIV disease. Subjects with HIV or without HIV infection who have no contraindications to lymph node biopsy will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
HIV persistence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States